CLINICAL TRIAL: NCT05913466
Title: Intraprostatic Injection of Tranexamic Acid Decrease Blood Loss During Monopolar TURP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tamer Abd El-Wahab Diab, Lecturer of Urology, Faculty of Medicine, Benha University, Benha, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Rc 5-5-2022
Record Dates: First submitted 2023-06-05; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Benign Prostatic Hyperplasia; Transurethral Resection of the Prostate; Tranexamic Acid
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid group (Experimental): Patients in this group will receive 1 gm of Tranexamic Acid (Cyklokapron) that will be dissolved in 50 ml of injectable 0.9% saline
  Interventions: Drug: Tranexamic Acid group
- Distilled water group (Placebo Comparator): This group will receive 10 mL of distilled water (placebo) in 1 L of irrigation solution sterile wash (glycine).
  Interventions: Drug: Distilled water group

INTERVENTIONS:
Drug: Tranexamic Acid group — Patients in this group will receive 1 gm of Tranexamic Acid (Cyklokapron) that will be dissolved in 50 ml of injectable 0.9% saline
  Arms: Tranexamic Acid group
Drug: Distilled water group — This group will receive 10 mL of distilled water (placebo) in 1 L of irrigation solution sterile wash (glycine).
  Arms: Distilled water group

SUMMARY:
This study aims to assess the role of intraprostatic injection of tranexamic acid in decreasing the blood loss during Transurethral resection of the prostate.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a process in which the pathology results in increased number of both stromal and epithelial cells in the area of the prostate around the urethra, which is pathologically known as hyperplasia, and not hypertrophy.

The accurate cause is not well known; however, "reactivation" of embryonic processes is one of the hypotheses that may cause benign prostatic hyperplasia (BPH). Benign prostatic hyperplasia (BPH) is a common condition that affects elderly men. Recently, many noninvasive and mini-invasive modalities have become popular for the management of men with voiding symptoms.

Transurethral resection of the prostate (TURP) is one of the most common and well-developed techniques used to treat benign prostatic hyperplasia (BPH), recognized as the 'gold standard' of the surgical treatments of enlarged prostates. The most relevant complications are the inability to void (5.8%), surgical revision (5.6%), urinary tract infection (UTI) (3.6%), bleeding requiring transfusions (2.9%), and Transurethral resection syndrome (1.4%). As the prostate has a rich blood supply, bleeding is one of the most common complications of Transurethral resection of the prostate.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an age between 50 and 85 years old
* who had benign prostatic hyperplasia (aged 50-85 years) with a prostate weight of 50-80 g.
* undergoing Transurethral resection of the prostate

Exclusion Criteria:

* Patient refusal.
* Patients hypersensitive to Tranexamic Acid, or on antiplatelet and anticoagulant drugs.
* Patients with a history of thrombotic events, bleeding disorders, chronic kidney disease.
* Patients with abnormal liver function test.
* Patients with cardiovascular disease and receiving with a drug-eluting stent, bladder stone, urethral stricture, or with previous prostate surgery, prostate cancer, with a UTI or who receiving 5α-reductase inhibitors.

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient with an age between 50 and 85 years old who had benign prostatic hyperplasia (aged 50-85 years) with a prostate weight of 50-80 g undergoing Transurethral resection of the prostate.
Enrollment: 60 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Amount of Blood Loss During Monopolar transurethral resection of the prostate | 2 weeks Postoperatively
  The efficacy of intraprostatic injection of tranexamic acid in reducing intraoperative bleeding will be assessed in litter.

SECONDARY OUTCOMES:
Hemoglobin (Hb) level | 2 weeks Postoperatively
  This outcome evaluates the changes in hemoglobin (Hb) level before and after the monopolar transurethral resection of the prostate (TURP) procedure.
Hematocrit (HCT) Level | 2 weeks Postoperatively
  This outcome evaluates the changes in hematocrit (HCT) level before and after the monopolar transurethral resection of the prostate (TURP) procedure.
Postoperative hospital stay length | 2 weeks Postoperatively
  Postoperative hospital stay length will be assessed in days

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be available under a clear request for the primary investigator
Supporting Information: Study Protocol
Time Frame: One year after the end of the trial

REFERENCES:
- [Derived] Diab T, El Hamshary SA, Abou Elezz A, El-Dakhakhny AS. Intraprostatic Injection of Tranexamic Acid Decrease Blood Loss During Monopolar Transurethral Resection of the Prostate: A Randomized Controlled Clinical Trial. Urology. 2024 Sep;191:119-126. doi: 10.1016/j.urology.2024.05.015. Epub 2024 May 22. PMID 38788904